CLINICAL TRIAL: NCT01228877
Title: The Effect of 16 Weeks of Hip Adduction and Abduction Resistance Exercise Training on Strength and Density of the Proximal Femur
Brief Title: The Effect of 16 Weeks of Hip Adduction and Abduction Resistance Exercise
Acronym: Ad/Ab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Space Biomedical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Ad/Ab exercise
Record Dates: First submitted 2010-10-08; First posted 2010-10-27 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Osteoporosis; Osteopenia; Sarcopenia
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Sarcopenia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): Adduction, Abduction and Squat exercise three times a week for 16 weeks
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Adduction, Abduction and Squat exercise three times a week for 16 weeks

SUMMARY:
Performing adduction and abduction resistance exercise will increase hip bone density and strength to a greater extent than doing squat and deadlift exercise.

Aim #1: To determine if doing hip adduction and abduction resistance exercise training for 16 weeks improves spine bone mineral density and hip bone mineral density and strength as determined by finite element modeling.

Aim #2: To compare the effects of hip adduction and abduction exercise to squat and deadlift exercise with respect to potential changes in hip bone mineral density and strength.

Aim #3: To determine if the addition of adduction and abduction exercise to squat and deadlift exercise promotes an "additive" effect with respect to changes in spine bone mineral density and hip bone mineral density and bone strength.

DETAILED DESCRIPTION:
The investigators will carry out a 16-week exercise training study (n=24) consisting of 3 groups (n=8 per group) of healthy, non-resistance trained adult men and women (age 25-55 years). Our aim is to determine if hip adduction and abduction resistance exercise is more effective than squat and deadlift exercise with respect to changes in the whole bone strength and density of the proximal femur and spine.

Group A will do only hip adduction and abduction exercises. Group B will do only squat and deadlift exercise Group C will do a combination of hip adduction and abduction and squat and deadlift exercise

Subjects will be imaged with quantitative computed tomography (QCT) of the proximal femur and spine, pre-training and post-training, to determine changes in spinal bone density and proximal femoral bone density and strength.

Serum assays of bone formation (osteocalcin) and bone resorption (serum CTX type I) will be performed four times during the study at 4 week intervals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Age of 25 to 55 years old

Exclusion Criteria:

* Hypertension (High blood pressure)
* Diabetes or metabolic syndrome
* Hyperlipidemia (High cholesterol)
* Cardiovascular Disease
* Asthma or other pulmonary disease (i.e. COPD)
* not pregnant
* have no joint or mobility limitations
* do not exercise on a regular basis

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2010-12; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Reduce risk of hip fracture | 16 weeks
  The investigators have prioritized the last year of NSBRI funding to test one the capabilities of our device, standing hip adduction/abduction exercise, to strengthen the proximal femoral bone. We believe that if we are able to detect increases in bone density and strength (assessed using quantitative computed tomography of the hip pre- and post-training) in healthy volunteers, this will be solid preliminary evidence to support modification of exercise protocols currently being used to reduce the rate of bone loss on the International Space Station.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lang, PhD, Principal Investigator — UCSF-Department of Radiology
Locations (1):
- UCSF-Department of radiology-China Basin, San Francisco, California, United States